CLINICAL TRIAL: NCT02240056
Title: Pilot Study: Central Nervous System and Hormonal Changes In Takotsubo Cardiomyopathy
Brief Title: Brain fMRT In Takotsubo Cardiomyopathy
Acronym: TAKINSULA
Status: Completed | Type: Observational
Sponsor: Wolfgang Dichtl, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Wolfgang Dichtl, MD PhD, Priv.Doz. DDr., Medical University Innsbruck
Organization: Medical University Innsbruck (Other)
Other Study IDs: TAKINSULA
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Takotsubo Cardiomyopathy
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- TTC: postmenopausal women with acute Takotsubo cardiomyopathy (TTC), diagnosis by coronary angiography within 24 hours of symptom onset
- NSTEMI / STEMI: postmenopausal women with acute ST elevation myocardial infarction (NSTEMI / STEMI), diagnosis by coronary angiography within 24 hours of symptom onset
- healthy subjects: healthy postmenopausal women without coronary artery disease

SUMMARY:
Certain cardiac and neurologic diseases influence each other via a still poorly understood "brain-heart axis". Subarachnoidal bleedings are well known to cause ECG alterations resembling those of myocardial infarction, along with a reduction of systolic myocardial function ("neurogenic stunned myocardium"). Alterations of the right insula region by a stroke or intracranial hemorrhage go along with a sympathetic activation (increased circulating catecholamine levels, tachycardia, arterial hypertension). In contrast, alterations of the left insula region often cause vagal reactions such as bradycardia, arterial hypotension. Takotsubo cardiomyopathy (TTC) is a just recently recognised subform of heart attacks, often caused by psychological or physical stress (death of a beloved one, divorce, job loss, infection, preoperative state). In more than 90% of cases, TTC affects postmenopausal women.

Functional MRT enables imaging of activated brain regions, either without ("resting state") or with specific stimuli. The investigators speculate that there is a specific involvement of the insula region during TTC.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal females aged below 90 years
* Informed written consent
* TTC or NSTEMI / STEMI undergoing coronary angiography within 24 hours of symptom onset

Exclusion Criteria:

* Delayed coronary angiography (> 24 hours after symptom onset)
* Inability to perform rsfMRT within the first 72 hours after coronary angiography
* Inability to communicate in German language
* Contraindications for a MRT examination (including pacemaker, implantable cardioverter-defibrillator, mechanical heart valves, claustrophobia, severe adipositas)
* Drug addiction, under guardianship
* Inability to stick to the follow up examination

Max Age: 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal women with TTC or NSTEMI / STEMI aged below 90 years
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Changes in brain functional MRT (resting state, paradigma) in postmenopausal females suffering from TTC as compared to NSTEMI / STEMI postmenopausal female patients | Within the first 72h after diagnosis and after 4-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Dichtl, MD PhD, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria